CLINICAL TRIAL: NCT00673283
Title: Early Detection of Lung Cancer Via Bi-plane Correlation Chest Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00008644; 2485-07-6R6
Record Dates: First submitted 2008-05-04; First posted 2008-05-07 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer; Metastatic Cancer in the Lungs
Keywords: lung cancer; nodules; radiography; CT; Stereoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: bi-plane chest radiography

INTERVENTIONS:
Device: bi-plane chest radiography — Bi-plane radiography of the thorax

SUMMARY:
This project proposes a new method, Bi-plane Correlation Imaging (BCI), for improved detection of subtle lung nodules. In BCI, two digital radiographs of the chest are acquired within a short time interval from slightly different posterior projections. The image data are incorporated into an enhanced Computer-aided Diagnosis (CAD) algorithm in which nodules present in the thoracic cavity are detected by examining the geometrical correlation of the detected signals in the two views. The data are alos viewed stereoscopically for visual diagnosis. The expected high sensitivity/specificity of the method has the potential to change the current state of practice, perhaps leading to a preventive lung cancer screening program for high-risk populations, similar to the mammography screening program currently in place for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Normal individuals
* Individuals with CT-confirmed subtle lung nodules.

Exclusion Criteria:

* Individuals with acute pulmonary abnormalities or those in poor health conditions will be excluded due to the potential impact on the results as well as difficulty of acquiring the images. Pregnant women will also be excluded to avoid the exposure of the fetus to radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The technique is effective in diagnosing early lung tumors. | end of the study

SECONDARY OUTCOMES:
The relative performance of BCI with respect to chest radiography and CT for lung cancer detection. | end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Samei, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medcal Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Samei E, Stebbins SA, Dobbins JT 3rd, McAdams HP, Lo JY. Multiprojection correlation imaging for improved detection of pulmonary nodules. AJR Am J Roentgenol. 2007 May;188(5):1239-45. doi: 10.2214/AJR.06.0843. PMID 17449766